CLINICAL TRIAL: NCT01930474
Title: Analysis of Mechanism of Resistance to Chemotherapy by Sequencing of Plasma DNA
Brief Title: Analysis of Plasma Tumor DNA in Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Chang, Assistant Professor, Seoul National University Hospital
Other Study IDs: 02-2013-105; B-1307/210-005 (Other: SeoulNUH)
Record Dates: First submitted 2013-08-21; First posted 2013-08-29 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Non Small Cell Lung Cancer Patients
Keywords: lung cancer, plasma DNA, free DNA, EGFR, ALK
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The presence of genetic alterations in the tyrosine kinase domain of the oncogene (eg. EGFR and ALK) is associated with the clinical response to tyrosine kinase inhibitors (TKIs) in patients with non-small cell lung cancers. Therefore, the detection of altered genetic alterations is useful for predicting the treatment response for TKIs in non-small cell lung cancer patients. However, good quality tumor tissues are available only in <50% of patients with inoperable lung cancer for mutation analysis. In this study, the investigators will detect and quantify the genetic alterations in plasma. the investigators will investigate if the serial measurement of cancer-derived genetic alterations in plasma can provide a means for monitoring disease progression, as well as treatment response. In addition the investigators will analysis the resistant mechanism of TKIs and chemotherapy with plasma tumor DNA.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically confirmed diagnosis of non-small cell lung cancer
* Have molecular evidence of genetic alterations in tumor sample (eg. EGFR mutations, ALK fusions)
* Patients must have given written informed consent

Exclusion Criteria:

* Patients who refuse the blood samplings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The non-small cell lung cancer patients who will be or have been treated with chemotherapy (including target agents)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Detection of genetic alterations (including EGFR and ALK) in plasma samples | 60 months
  To evaluate the sensitivity of digital PCR to detect the genetic alterations in plasma tumor DNA

SECONDARY OUTCOMES:
Quantifying circulating tumor DNA in serially collected plasma specimens | 60 months
  To evaluate the change of quantity of circulating tumor DNA with digital PCR

OTHER OUTCOMES:
Analysis of genetic alterations related with drug-resistance with next generation genome sequencing | 24 months
  The tumor DNA will be sequenced and analyzed with NGS to detect the genetic alterations related with drug-resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Chang, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea